CLINICAL TRIAL: NCT01212783
Title: Treatment of Maternal Depression in Home Visitation: Mother and Child Impacts
Acronym: MIDISII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH087499-01A1 (NIH)
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Depressive Disorder in Mothers
Keywords: depression; psychological treatments; Cognitive Behavioral Therapy; child development; parenting; home visitation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Present-Centered Therapy (Active Comparator): Mothers will receive 15 weekly sessions of PCT plus two monthly booster sessions following the 15th session.
  Interventions: Behavioral: Present-Centered Therapy
- In-Home Cognitive Behavioral Therapy (Experimental): Mothers will receive 15 weekly sessions of IH-CBT plus two booster sessions scheduled monthly following the 15th session.
  Interventions: Behavioral: In-Home Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: In-Home Cognitive Behavioral Therapy — Adapted form of CBT that is delivered in the home setting, uniquely designed for young, low income new mothers, and is explicitly integrated with home visitation. IH-CBT is delivered by a masters level therapist. It consists of 15 weekly sessions and two monthly booster sessions provided after the 15th session.
  Arms: In-Home Cognitive Behavioral Therapy
Behavioral: Present-Centered Therapy — Present-Centered Therapy is a supportive psychotherapy.
  Arms: Present-Centered Therapy

SUMMARY:
The purpose of this study is to determine the efficacy of In-Home Cognitive Behavioral Therapy (IH-CBT) in comparison to Present-Centered Therapy (PCT), a supportive therapeutic approach. IH-CBT is adapted form of CBT that is provided to depressed mothers participating in ongoing home visitation services. IH-CBT has been adapted to fit the setting, population, and context associated with home visiting. Mothers are recruited at 4 months postpartum. A comprehensive assessment battery is administered at pre-treatment, post-treatment, and 6, 12, and 18 months after the end of treatment. It is hypothesized that IH-CBT will be superior to PCT in decreasing depression, improving overall functioning, enhancing parenting effectiveness, and preventing relapse.

DETAILED DESCRIPTION:
Home visitation is a prevention program for sociodemographically high risk, first-time mothers and their children that is designed to optimize maternal life course and child trajectories. Research indicates that maternal depression (1) is a significant problem in home visitation with up to 45% of mothers experiencing clinically elevated symptoms while only 14% receive treatment, and (2) can significantly interfere with the efficacy of home visitation. Moreover, maternal depression negatively impacts mother-child interactions and child functioning thus potentially precluding the dyad from fully benefiting from home visitation. To address the high rate of maternal depression in existing home visitation programs, In-Home Cognitive Behavior Therapy (IH-CBT) was developed through an R34 grant as a treatment for mothers in home visitation experiencing depression postpartum. IH-CBT consists of the core features of CBT that have been adapted to address the unique needs and challenges of mothers receiving home visitation. Findings from the R34 indicate that IH-CBT is highly effective at reducing depression, with 66.7% of depressed mothers no longer obtaining a diagnosis of MDD at the end of treatment in contrast to a rate of 24.3% in mothers receiving home visitation alone. In addition, mothers receiving IH-CBT reported increased social support and reduction in other psychiatric symptoms, much of which was maintained at 3 month follow-up. This study seeks to replicate IH-CBT with a larger sample, compare the treatment to a more rigorous control condition (Present-Centered Therapy-PCT), and extend follow-up to 18 months in order to determine relapse rate. There is mixed evidence regarding the long-term effectiveness of home visitation on depressed mothers and their children-critical outcomes that, if adequately demonstrated, would significantly enhance the public health implications of home visitation. Accordingly, the study also seeks to examine the impact of IH-CBT and recovery from depression on parenting and children. Specifically, 220 mothers who are enrolled in home visitation will be recruited through initial screening and subsequent diagnosis of MDD. Subjects will be randomly assigned to IH-CBT + home visitation or PCT + home visitation. Both IH-CBT and PCT will be implemented in 15 sessions with two booster sessions provided 1 and 2 months after treatment. Measures of depression, psychiatric comorbidity, adaptive functioning, social support, parenting, and child functioning will be administered at pre-treatment, post-treatment, and at 6, 12 and 18 month follow-ups after post-treatment. It is hypothesized that IH-CBT will be superior to PCT in (1) recovery from depression, (2) risk of relapse and recurrence, and (3) increasing social support and reducing overall psychiatric symptomatology. In addition, mothers who recover from depression will show improvements in parenting and the mother-child relationship, and their children will achieve improved cognitive, social, emotional, and biologic outcomes, relative to non-recovered mothers and their offspring.

ELIGIBILITY:
Inclusion Criteria:

* first-time mother participating in home visitation program
* enrolled in home visitation program for at least 2 months
* 16 years of age or older
* score of 11 or higher on Edinburgh Perinatal Depression Screen at 3 months postpartum
* diagnosis of Major Depressive Disorder using SCID
* English speaking

Exclusion Criteria:

* lifetime history of bipolar disorder, schizophrenia, mental retardation, organic brain syndrome, antisocial personality disorder
* history of psychosis
* current substance dependence
* current antidepressant use or other mood altering medications and/or current involvement in psychotherapy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
maternal depression | 23 months
  Maternal depression as measured by self-report, clinician rating based on semi-structured interview, and psychiatric diagnosis based on semi-structured interview.

SECONDARY OUTCOMES:
child development and social/emotional functioning | 23 months
  Child developmental status based on standardized developmental assessment, and maternal report of child social/emotional functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Robert T. Ammerman, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States